CLINICAL TRIAL: NCT04326660
Title: The Smartphone-Based Cancer and Obesity Prevention Education Program for Chinese Women (SCOPE-Chinese Women)
Brief Title: SCOPE-Chinese Women Study
Acronym: SCOPE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Central South University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 18-27025; 217516 (Other: University of California, San Francisco)
Record Dates: First submitted 2020-03-23; First posted 2020-03-30 (Actual); Last update posted 2022-12-22 (Actual); Status verified 2022-12

CONDITIONS: Cancer, Breast; Obesity, Abdominal
Keywords: Obesity; Abdominal; Cancer Prevention
MeSH Terms: conditions — Breast Neoplasms; Obesity, Abdominal; Obesity

STUDY DESIGN:
Intervention Model Description: This pilot study will utilize a randomized control trail design with a control group.
Who Masked: Participant
Masking Description: To decrease cross-contamination of treatment effect, the six study sites will be the units of randomization. A Statistical Package for Social Sciences (SPSS) program will be used to statistically match the groups and to randomly assign each study group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): Participants in the control group will receive a Fitbit Alta-Heart Rate (HR) and 12 weekly non-tailored educational modules via WeChat on general health topics that are important to 20-45 year-old women in China. Topics include intimate partner violence, anxiety, depression, sexually transmitted infections, HIV, unintended pregnancy, hepatitis B, and general cancer prevention.
- SCOPE-Chinese Women Intervention (Experimental): SCOPE-Chinese Women intervention content and methods: SCOPE-Chinese Women is a smartphone- based intervention.
  Component 1. All study participants will receive a Fitbit Alta-HR tracking device to wear daily. Each participant will receive in-person, training on how to access the app and their tracking data. If a participant has not used the fitness device and app for more than one week, a WeChat reminder message will be sent to the participant.
  Component 2. Participants will receive 12 weekly culturally appropriate and evidence-based SCOPE-Chinese Women educational modules along with tailored tips and messages via WeChat. Each module will include three educational sessions that last less than 45 minutes total.
  Component 3. Six bi-weekly messages will be sent to participants via WeChat to encourage positive behavioral changes. Each participant's message content will be based on the participant's tracker information, personal goals, and preferences.
  Interventions: Other: SCOPE-Chinese Women

INTERVENTIONS:
Other: SCOPE-Chinese Women — SCOPE-Chinese Women is a smart-phone based intervention that includes a Fitbit tracking device to monitor daily activity, 12-weeks of educational modules delivered by WeChat, and Bi-weekly messages that encourage positive behavioral change. The data will be examined by the research team to assess efficacy of the intervention.
  Arms: SCOPE-Chinese Women Intervention

SUMMARY:
This project examines the feasibility of a smartphone-based intervention to reduce obesity and breast cancer risk among Chinese women in China. The proposed intervention is to use the mobile application and an activity tracker device to promote a healthier lifestyle and physical activity. The intervention will be tailored to the participants' behaviors, personal needs, and preferences. The aim is to reduce abdominal obesity and improve healthy lifestyle behaviors in premenopausal women with children in order to reduce the growing cancer burden in China.

DETAILED DESCRIPTION:
Cancer presents a major disease burden across the globe. The incidence and mortality of gynecologic cancers have increased significantly in China over the last two decades with breast and endometrial cancer as leading causes of death in women in China. Obesity, especially abdominal obesity, and unhealthy lifestyles are major risk factors for breast and endometrial cancer. A high risk group for obesity is mothers with dependent children as they have high levels of stress and family responsibilities that prevent regular engagement in a healthy lifestyle and early screening activities. Because reducing postmenopausal abdominal obesity is very difficult and because of the significant increased risk for gynecologic cancers in obese postmenopausal women, interventions that aim to reduce abdominal obesity and improve healthy lifestyle behaviors in premenopausal women with children are critical to reducing the growing cancer burden in China. A smartphone-based intervention provides a promising platform for obesity and cancer prevention. In this proposed study, the research team will modify the Healthy Mothers Healthy Children: Technology-Based Intervention to Prevent Obesity, which was developed by the principal investigator. The proposed intervention (titled "The Smartphone-Based Cancer and Obesity Prevention Education Program for Chinese Women: SCOPE-Chinese Women") is a smartphone-based, data-driven, and individually tailored intervention. It includes 12 weekly educational modules and six bi-weekly tailored messages delivered via WeChat, a popular communication app in China. The intervention will also be tailored to the participants' behaviors, personal needs, and preferences. The overall goal of this proposed study is to assess the feasibility and estimate the preliminary efficacy of the SCOPE-Chinese Women intervention using a randomized control study design (RCT). The following aims will be addressed.

Aim 1: To assess the feasibility of the smartphone-based lifestyle intervention (i.e., SCOPE-Chinese Women).

Aim 2: To estimate the preliminary efficacy of the SCOPE-Chinese Women intervention on the primary outcome (waist circumference) and secondary outcomes (body mass index, self-efficacy, food intake, physical activity, and metabolic risk) between the intervention and control groups at baseline, 3 months, and 6 months.

Aim 3: To understand participants' acceptance, barriers to adherence, and recommendations for intervention.

ELIGIBILITY:
Inclusion Criteria:

Participants must:

* Be female
* Be at least 18 years old
* Have a waist circumference great than 80 cm
* Own a smartphone
* Be able to read Chinese and speak Mandarin
* Be premenopausal
* Have a child between the age of 1 and 18 years old

Exclusion Criteria:

Women are excluded from the study if they:

* Are pregnant
* Gave birth less than 12 months prior to enrollment date
* Have an acute or life-threatening disease (e.g., renal failure).

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2020-07-20 (Actual); Primary Completion 2021-12-30 (Actual); Study Completion 2021-12-30 (Actual)

PRIMARY OUTCOMES:
Mean Change in Waist Circumference Over Time | Baseline, 3 months, and 6 months
  The National Institutes of Health (NIH) waist circumference measurement protocol will be used to measure change in waist circumference for each participant over time.

SECONDARY OUTCOMES:
Mean Change in Body Mass Index (BMI) Over Time | Baseline, 3 months, and 6 months
  Weight and height will be used to compute the BMI with the formula=weight (kilograms(kg)) / height in (meters squared (m2). Changes in BMI will be collected for each participant over time.
Mean Change in Scores on the Self-Rated Abilities for Health Practices Scale Over Time | Baseline, 3 months, and 6 months
  The Self Rated Abilities for Health Practices Scale (SRAHP) is a 28-item survey, with each item scored on a 5-point scale, with item scores ranging from 0=Not at all to 4=Completely. The survey is designed to measure self-perceived ability to implement health-promoting behaviors across four subscales: Exercise, Nutrition, Responsible Health Practice, and Psychological Well Being, and overall. The total score ranges from 0 - 112, with higher scores indicating greater abilities for health practices. Changes in scores will be collected for each participant over time.
Mean Changes in China Food Frequency Questionnaire (FFQ) over time. | Baseline, 3 months, and 6 months
  Food intake using the China food frequency questionnaire (FFQ), which includes a list of 118 food items will be used to measure aggregate changes in food intake over time.
Mean Changes in Overall Physical Activity | Baseline, 3 months, and 6 months
  Change in overall Physical activity over time will be measured using the Fitbit Alta-HR device for 10 hours while participants are awake.
Mean Change in Blood Pressure Over Time | Baseline, 3 months, and 6 months
  Changes in blood pressure will be measured using the YuWell YE690A monitor for each participant over time.
Mean Change in Hemoglobin A1C (HbA1C) Over Time | Baseline and 6 months
  A blood sample will be collected to measure change in HbA1C over time for each participant, using an established cut off value at 6.4%.
Mean Change in Serum Lipid Levels Over Time | Baseline and 6 months
  A blood sample will be collected to measure change in total cholesterol, low-density lipoprotein (LDL) cholesterol, high-density lipoprotein (HDL) cholesterol, and triglycerides (all measured in milligrams per deciliter (mg/dL)) over time for each participant
Mean Change in Cortisol over time | Baseline and 6 months
  A blood sample will be collected to measure change in total cortisol levels over time for each participant.

OTHER OUTCOMES:
Percentage of Eligible participants Who Agree To Be Screened | At Baseline
  The number of overall eligible participants and the number of eligible participants who agree to be screened will be used to compute the percentage used for enrollment.
Number of Uses of The Tracking App Over Time | Baseline to 6 months
  The number of uses of the tracking app and frequency of accessing the 12 modules, to measure change in usability over time
Percentage of Participants who completed assessments | Up to 6 months
  The percentage of completed assessments by participants at each visit will be used to measure adherence over time

CONTACTS AND LOCATIONS:
Overall Officials: Jyu-Lin Chen, RN, PhD, Principal Investigator — University of California, San Francisco; Jia Guo, RN, PhD, Principal Investigator — Central South Univeristy
Locations (2):
- University of California, San Francisco, San Francisco, California, United States
- Central South University, Yuelucun, Changsha, Hunan, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fan L, Strasser-Weippl K, Li JJ, St Louis J, Finkelstein DM, Yu KD, Chen WQ, Shao ZM, Goss PE. Breast cancer in China. Lancet Oncol. 2014 Jun;15(7):e279-89. doi: 10.1016/S1470-2045(13)70567-9. PMID 24872111
- [Background] Jiang X, Tang H, Chen T. Epidemiology of gynecologic cancers in China. J Gynecol Oncol. 2018 Jan;29(1):e7. doi: 10.3802/jgo.2018.29.e7. PMID 29185265
- [Background] Fair AM, Dai Q, Shu XO, Matthews CE, Yu H, Jin F, Gao YT, Zheng W. Energy balance, insulin resistance biomarkers, and breast cancer risk. Cancer Detect Prev. 2007;31(3):214-9. doi: 10.1016/j.cdp.2007.04.003. Epub 2007 Jul 23. PMID 17646056
- [Background] Wang X, Li L, Gao J, Liu J, Guo M, Liu L, Wang W, Wang J, Xing Z, Yu Z, Wang X. The Association Between Body Size and Breast Cancer in Han Women in Northern and Eastern China. Oncologist. 2016 Nov;21(11):1362-1368. doi: 10.1634/theoncologist.2016-0147. Epub 2016 Aug 5. PMID 27496041
- [Background] Cutrona CE, Abraham WT, Russell DW, Beach SR, Gibbons FX, Gerrard M, Monick M, Philibert R. Financial strain, inflammatory factors, and haemoglobin A1c levels in African American women. Br J Health Psychol. 2015 Sep;20(3):662-79. doi: 10.1111/bjhp.12120. Epub 2014 Oct 18. PMID 25327694
- [Background] Landstedt E, Harryson L, Hammarstrom A. Changing housework, changing health? A longitudinal analysis of how changes in housework are associated with functional somatic symptoms. Int J Circumpolar Health. 2016 Jun 30;75:31781. doi: 10.3402/ijch.v75.31781. eCollection 2016. PMID 27369590
- [Background] Berge JM, Larson N, Bauer KW, Neumark-Sztainer D. Are parents of young children practicing healthy nutrition and physical activity behaviors? Pediatrics. 2011 May;127(5):881-7. doi: 10.1542/peds.2010-3218. Epub 2011 Apr 11. PMID 21482603
- [Background] Liu Y, Warren Andersen S, Wen W, Gao YT, Lan Q, Rothman N, Ji BT, Yang G, Xiang YB, Shu XO, Zheng W. Prospective cohort study of general and central obesity, weight change trajectory and risk of major cancers among Chinese women. Int J Cancer. 2016 Oct 1;139(7):1461-70. doi: 10.1002/ijc.30187. Epub 2016 May 31. PMID 27177094
- [Background] Sun A, Cheng J, Bui Q, Liang Y, Ng T, Chen JL. Home-Based and Technology-Centered Childhood Obesity Prevention for Chinese Mothers With Preschool-Aged Children. J Transcult Nurs. 2017 Nov;28(6):616-624. doi: 10.1177/1043659617719139. Epub 2017 Jul 8. PMID 28826348
- [Background] Guan X, Sun G, Zheng L, Hu W, Li W, Sun Y. Associations between metabolic risk factors and body mass index, waist circumference, waist-to-height ratio and waist-to-hip ratio in a Chinese rural population. J Diabetes Investig. 2016 Jul;7(4):601-6. doi: 10.1111/jdi.12442. Epub 2015 Dec 26. PMID 27181937
- [Background] Wen X, Mai J, Gao X, Guo M, Wu Y, Liu X, Zhao L. [Cut-off values of waist circumference for central obesity in Chinese adults]. Zhonghua Xin Xue Guan Bing Za Zhi. 2015 Sep;43(9):822-6. Chinese. PMID 26652826
- [Background] Nanayakkara J, Lekamwasam S. Validity of BMI, hip and waist circumferences as surrogate measures of obesity in a cohort of Sri Lankan premenopausal women. Ceylon Med J. 2013 Jun;58(2):72-5. doi: 10.4038/cmj.v58i2.4720. PMID 23817937
- [Background] Singhal N, Mathur P, Pathak R. Validity of simple, novel measures of generalized and central obesity among young Asian Indian women. Indian J Med Sci. 2011 Dec;65(12):518-27. PMID 23548252
- [Background] Yu R, Yan LL, Wang H, Ke L, Yang Z, Gong E, Guo H, Liu J, Gu Y, Wu Y. Effectiveness of a community-based individualized lifestyle intervention among older adults with diabetes and hypertension, Tianjin, China, 2008-2009. Prev Chronic Dis. 2014 May 15;11:E84. doi: 10.5888/pcd11.120333. PMID 24831288
- [Background] Zhang R, Li Y, Zhang S, Cai X, Zhou X, Ji L. The Association of Retinopathy and Plasma Glucose and HbA1c: A Validation of Diabetes Diagnostic Criteria in a Chinese Population. J Diabetes Res. 2016;2016:4034129. doi: 10.1155/2016/4034129. Epub 2016 Oct 11. PMID 27807545